CLINICAL TRIAL: NCT07032870
Title: Pilot Study: Validation of Operators and Inter-Evaluator Variability in Diagnostic Strategies for ICU-Acquired Weakness (NMusICU-R)
Brief Title: Physical Therapist Inter-Rater Reliability in Neuro-Muscle Ultrasound in Critically Ill Patients
Acronym: NMusICU-R
Status: Recruiting | Type: Observational
Sponsor: University of Chile (Other)
Collaborators: Clinica Indisa (Other)
Responsible Party: Principal Investigator, Oscar Arellano, PhD. Candidate in Biomedical Sciences, University of Chile
Other Study IDs: 176-25-24
Record Dates: First submitted 2025-06-11; First posted 2025-06-24 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Critical Illness
Keywords: critical illness; ultrasound; Inter-rater reliability; physical therapist
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically Ill Patients: Adult ICU patients at Clínica INDISA evaluated by three physical therapists using bedside ultrasound of the quadriceps muscle and peripheral nerves, and assessed with clinical scales (MRC-SS and FSS-ICU) to measure inter-rater reliability and correlation of results.

SUMMARY:
The goal of this observational study is to evaluate the feasibility and inter-rater reliability of muscle and peripheral nerve ultrasound for the early detection of ICU-acquired weakness (ICU-AW) in critically ill patients.

The main questions it aims to answer are:

Can ICU physical therapists consistently measure muscle and nerve ultrasound variables such as muscle thickness, cross-sectional area, pennation angle, and echogenicity in critically ill patients?

Do clinical scales (MRC-SS and FSS-ICU) show inter-evaluator agreement and correlate with ultrasound findings?

Participants are adult ICU patients at Clínica INDISA who are undergoing routine neuromuscular assessments by trained physical therapists. Each patient will be evaluated by three independent raters using ultrasound and standardized clinical scales. Data will be collected and analyzed to determine inter-rater reliability and correlations between clinical and imaging findings.

DETAILED DESCRIPTION:
This observational, cross-sectional pilot study aims to assess the inter-rater reliability of muscle and peripheral nerve ultrasound and functional clinical scales in the diagnosis of ICU-acquired weakness (ICU-AW). The study involves adult patients admitted to the Adult Critical Care Unit at Clínica INDISA (Santiago, Chile). Participants will undergo muscle ultrasound of the quadriceps (measuring anterior compartment thickness, cross-sectional area, and pennation angle) and peripheral nerve ultrasound (assessing cross-sectional area and echogenicity of specific nerves) performed by three trained physical therapists. Clinical assessments using the MRC Sum Score (MRC-SS) and the Functional Status Score for the ICU (FSS-ICU) will also be performed by each rater.

The main aim is to evaluate the agreement between raters using the intraclass correlation coefficient (ICC) for ultrasound variables and Kendall's W for functional scales. The study will also explore correlations between clinical scores and ultrasound findings using Pearson or Spearman correlation coefficients. Echogenicity will be quantified using ImageJ software.

All procedures are performed at bedside using portable ultrasound equipment, and evaluations follow safety guidelines for critically ill patients. The results of this study will contribute to validating physical therapists as reliable operators for early identification of ICU-AW using ultrasound-based tools and standardized clinical assessments.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old) admitted to the Adult Intensive Care Unit (ICU) of Clínica INDISA.
* Conscious and clinically stable at the time of assessment.
* Able to provide written informed consent.

Exclusion Criteria:

* Known allergy to ultrasound gel.
* Body mass index (BMI) ≥ 30 kg/m².
* Pre-existing neuromuscular disease.
* Continuous renal replacement therapy or severe hepatic coagulopathy.
* Platelet count < 20,000/µL.
* Lower limb amputation or recent fractures.
* Ongoing chemotherapy or immunosuppressive treatment with corticosteroids.
* Epileptic status or pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients admitted to the Adult Intensive Care Unit (ICU) of Clínica INDISA in Santiago, Chile. Participants will be selected during their hospitalization for critical illness and evaluated on a randomly chosen day during their ICU stay. All participants will be physically and cognitively able to provide informed consent.
Sampling Method: Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2025-02-08 (Actual); Primary Completion 2025-12-09 (Estimated); Study Completion 2025-12-09 (Estimated)

PRIMARY OUTCOMES:
Inter-rater reliability of quadriceps muscle ultrasound measurements | Assessed once within 60 days following ICU admission
  Intraclass correlation coefficient (ICC) between three evaluators for ultrasound variables including quadriceps muscle thickness, rectus femoris and vastus intermedius cross-sectional area, and pennation angle.
Peripheral Nerve Ultrasound Inter-Rater Reliability | Assessed once within 60 days following ICU admission
  Intraclass correlation coefficient (ICC) between three evaluators for cross-sectional area and echogenicity of peripheral nerves (median, ulnar, tibial, and fibular) measured by ultrasound.

SECONDARY OUTCOMES:
Inter-rater agreement of Functional Status Score for the ICU (FSS-ICU) | Assessed once within 60 days following ICU admission
  Kendall's W coefficient to assess the level of agreement among three physical therapists applying the FSS-ICU scale in critically ill patients.
Inter-Rater Agreement of MRC Sum Score | Assessed once within 60 days following ICU admission
  Kendall's W coefficient to determine the agreement between three physical therapists applying the MRC-SS to assess muscle strength in ICU patients.
Correlation between clinical scales and ultrasound findings | Assessed once within 60 days following ICU admission
  Pearson or Spearman correlation coefficients between MRC-SS/FSS-ICU results and quantitative ultrasound parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Paola A Llanos, PhD, Study Chair — University of Chile
Locations (1):
- Clínica INDISA, Santiago, Metropolitan Region, Chile

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and legal restrictions. Only aggregate results derived from the analysis of anonymized data will be published in scientific articles. This decision follows the confidentiality agreements established in the informed consent and the approval granted by the institutional ethics committee.

REFERENCES:
- [Background] Lefaucheur JP, Nordine T, Rodriguez P, Brochard L. Origin of ICU acquired paresis determined by direct muscle stimulation. J Neurol Neurosurg Psychiatry. 2006 Apr;77(4):500-6. doi: 10.1136/jnnp.2005.070813. Epub 2005 Nov 23. PMID 16306155
- [Background] Formenti P, Umbrello M, Coppola S, Froio S, Chiumello D. Clinical review: peripheral muscular ultrasound in the ICU. Ann Intensive Care. 2019 May 17;9(1):57. doi: 10.1186/s13613-019-0531-x. PMID 31101987
- [Background] Paolo F, Valentina G, Silvia C, Tommaso P, Elena C, Martin D, Marini John J, Davide C. The possible predictive value of muscle ultrasound in the diagnosis of ICUAW in long-term critically ill patients. J Crit Care. 2022 Oct;71:154104. doi: 10.1016/j.jcrc.2022.154104. Epub 2022 Jul 4. PMID 35797827
- [Background] Lad H, Saumur TM, Herridge MS, Dos Santos CC, Mathur S, Batt J, Gilbert PM. Intensive Care Unit-Acquired Weakness: Not just Another Muscle Atrophying Condition. Int J Mol Sci. 2020 Oct 22;21(21):7840. doi: 10.3390/ijms21217840. PMID 33105809
- [Background] Elkalawy H, Sekhar P, Abosena W. Early detection and assessment of intensive care unit-acquired weakness: a comprehensive review. Acute Crit Care. 2023 Nov;38(4):409-424. doi: 10.4266/acc.2023.00703. Epub 2023 Nov 30. PMID 38052508
- [Background] Rajagopal K, Vijayan D, Thomas SM. Association of SOFA Score with Severity of Muscle Wasting in Critically Ill Patients: A Prospective Observational Study. Indian J Crit Care Med. 2023 Oct;27(10):743-747. doi: 10.5005/jp-journals-10071-24540. PMID 37908434
- [Background] Beekman R, Visser LH. High-resolution sonography of the peripheral nervous system -- a review of the literature. Eur J Neurol. 2004 May;11(5):305-14. doi: 10.1111/j.1468-1331.2004.00773.x. PMID 15142223
- [Background] Gruber L, Loizides A, Gruber H, Skalla E, Haushammer S, Horlings C, Beer R, Helbok R, Loscher WN. Differentiation of Critical Illness Myopathy and Critical Illness Neuropathy Using Nerve Ultrasonography. J Clin Neurophysiol. 2023 Nov 1;40(7):600-607. doi: 10.1097/WNP.0000000000000922. Epub 2022 Jan 25. PMID 35089907
- [Background] Grimm A, Decard BF, Axer H, Fuhr P. The Ultrasound pattern sum score - UPSS. A new method to differentiate acute and subacute neuropathies using ultrasound of the peripheral nerves. Clin Neurophysiol. 2015 Nov;126(11):2216-25. doi: 10.1016/j.clinph.2015.01.011. Epub 2015 Feb 3. PMID 25691156
- [Background] Hadda V, Khilnani GC, Kumar R, Dhunguna A, Mittal S, Khan MA, Madan K, Mohan A, Guleria R. Intra- and Inter-observer Reliability of Quadriceps Muscle Thickness Measured with Bedside Ultrasonography by Critical Care Physicians. Indian J Crit Care Med. 2017 Jul;21(7):448-452. doi: 10.4103/ijccm.IJCCM_426_16. PMID 28808365
- [Background] Di Matteo A, Moscioni E, Lommano MG, Cipolletta E, Smerilli G, Farah S, Airoldi C, Aydin SZ, Becciolini A, Bonfiglioli K, Carotti M, Carrara G, Cazenave T, Corradini D, Cosatti MA, de Agustin JJ, Destro Castaniti GM, Di Carlo M, Di Donato E, Di Geso L, Elliott A, Fodor D, Francioso F, Gabba A, Hernandez-Diaz C, Horvath R, Hurnakova J, Jesus D, Marin J, Martire MV, Mashadi Mirza R, Massarotti M, Musca AA, Nair J, Okano T, Papalopoulos I, Rosa J, Rosemffet M, Rovisco J, Rozza D, Salaffi F, Scioscia C, Scire CA, Tamas MM, Tanimura S, Ventura-Rios L, Villota-Eraso C, Villota O, Voulgari PV, Vreju FA, Vukatana G, Hereter JZ, Zanetti A, Grassi W, Filippucci E. Reliability assessment of ultrasound muscle echogenicity in patients with rheumatic diseases: Results of a multicenter international web-based study. Front Med (Lausanne). 2023 Jan 17;9:1090468. doi: 10.3389/fmed.2022.1090468. eCollection 2022. PMID 36733934
- [Background] Pardo E, El Behi H, Boizeau P, Verdonk F, Alberti C, Lescot T. Reliability of ultrasound measurements of quadriceps muscle thickness in critically ill patients. BMC Anesthesiol. 2018 Dec 27;18(1):205. doi: 10.1186/s12871-018-0647-9. PMID 30591032
- [Background] Karapinar M, Atilla Ayyildiz V, Unal M, Firat T. Ultrasound imaging of quadriceps muscle in patients with knee osteoarthritis: The test-retest and inter-rater reliability and concurrent validity of echo intensity measurement. Musculoskelet Sci Pract. 2021 Dec;56:102453. doi: 10.1016/j.msksp.2021.102453. Epub 2021 Sep 1. PMID 34507044
- [Background] Turan Z, Topaloglu M, Ozyemisci Taskiran O. Medical Research Council-sumscore: a tool for evaluating muscle weakness in patients with post-intensive care syndrome. Crit Care. 2020 Sep 18;24(1):562. doi: 10.1186/s13054-020-03282-x. No abstract available. PMID 32948221
- [Background] Derde S, Hermans G, Derese I, Guiza F, Hedstrom Y, Wouters PJ, Bruyninckx F, D'Hoore A, Larsson L, Van den Berghe G, Vanhorebeek I. Muscle atrophy and preferential loss of myosin in prolonged critically ill patients. Crit Care Med. 2012 Jan;40(1):79-89. doi: 10.1097/CCM.0b013e31822d7c18. PMID 21926599
- [Background] Wilcox SR. Corticosteroids and neuromuscular blockers in development of critical illness neuromuscular abnormalities: A historical review. J Crit Care. 2017 Feb;37:149-155. doi: 10.1016/j.jcrc.2016.09.018. Epub 2016 Sep 26. PMID 27736708
- [Background] Stevens RD, Marshall SA, Cornblath DR, Hoke A, Needham DM, de Jonghe B, Ali NA, Sharshar T. A framework for diagnosing and classifying intensive care unit-acquired weakness. Crit Care Med. 2009 Oct;37(10 Suppl):S299-308. doi: 10.1097/CCM.0b013e3181b6ef67. PMID 20046114
- [Background] Fan E, Cheek F, Chlan L, Gosselink R, Hart N, Herridge MS, Hopkins RO, Hough CL, Kress JP, Latronico N, Moss M, Needham DM, Rich MM, Stevens RD, Wilson KC, Winkelman C, Zochodne DW, Ali NA; ATS Committee on ICU-acquired Weakness in Adults; American Thoracic Society. An official American Thoracic Society Clinical Practice guideline: the diagnosis of intensive care unit-acquired weakness in adults. Am J Respir Crit Care Med. 2014 Dec 15;190(12):1437-46. doi: 10.1164/rccm.201411-2011ST. PMID 25496103
- [Background] Barreiro E. Models of disuse muscle atrophy: therapeutic implications in critically ill patients. Ann Transl Med. 2018 Jan;6(2):29. doi: 10.21037/atm.2017.12.12. PMID 29430446
- [Background] Wang W, Xu C, Ma X, Zhang X, Xie P. Intensive Care Unit-Acquired Weakness: A Review of Recent Progress With a Look Toward the Future. Front Med (Lausanne). 2020 Nov 23;7:559789. doi: 10.3389/fmed.2020.559789. eCollection 2020. PMID 33330523
- [Background] Schefold JC, Wollersheim T, Grunow JJ, Luedi MM, Z'Graggen WJ, Weber-Carstens S. Muscular weakness and muscle wasting in the critically ill. J Cachexia Sarcopenia Muscle. 2020 Dec;11(6):1399-1412. doi: 10.1002/jcsm.12620. Epub 2020 Sep 7. PMID 32893974
- [Background] Kress JP, Hall JB. ICU-acquired weakness and recovery from critical illness. N Engl J Med. 2014 Apr 24;370(17):1626-35. doi: 10.1056/NEJMra1209390. No abstract available. PMID 24758618
- [Background] Vanhorebeek I, Latronico N, Van den Berghe G. ICU-acquired weakness. Intensive Care Med. 2020 Apr;46(4):637-653. doi: 10.1007/s00134-020-05944-4. Epub 2020 Feb 19. PMID 32076765
- [Background] De Jonghe B, Sharshar T, Lefaucheur JP, Authier FJ, Durand-Zaleski I, Boussarsar M, Cerf C, Renaud E, Mesrati F, Carlet J, Raphael JC, Outin H, Bastuji-Garin S; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Paresis acquired in the intensive care unit: a prospective multicenter study. JAMA. 2002 Dec 11;288(22):2859-67. doi: 10.1001/jama.288.22.2859. PMID 12472328

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-08): https://cdn.clinicaltrials.gov/large-docs/70/NCT07032870/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-08): https://cdn.clinicaltrials.gov/large-docs/70/NCT07032870/ICF_001.pdf